CLINICAL TRIAL: NCT03148262
Title: Use of High-Flow Nasal Cannula to Prevent Desaturation Episodes in the Morbidly Obese Patients Undergoing Colonoscopy:A Prospective Randomized Clinical Trial
Brief Title: High-Flow Nasal Cannula and Desaturation Episodes in the Morbidly Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Christina Riccio, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU 112016-058
Record Dates: First submitted 2017-05-08; First posted 2017-05-10 (Actual); Results first posted 2018-11-19 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Desaturation of Blood; Obesity; Colonoscopy; Sleep Apnea; High Flow Nasal Cannula
MeSH Terms: conditions — Obesity; Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- The high flow nasal cannula (Experimental): The Comfort Flo system will be used for the high flow nasal cannula during colonoscopy
  Interventions: Device: The Comfort Flo system
- The standard nasal cannula (Placebo Comparator): The Salter nasal cannula will be used during the colonoscopy
  Interventions: Device: The Salter nasal cannula

INTERVENTIONS:
Device: The Comfort Flo system — The Comfort Flo system will be used for the high flow nasal cannula during procedural sedation
  Other Names: High flow nasal cannula
  Arms: The high flow nasal cannula
Device: The Salter nasal cannula — A Salter nasal cannula will be used at 4L/ minute during the procedural sedation.
  Other Names: Standard nasal cannula
  Arms: The standard nasal cannula

SUMMARY:
It is standard practice in the United States and many parts of world to perform Gastrointestinal (GI) endoscopy with the patient under deep sedation. Obesity is accepted as a patient specific risk factor for hypoxic events during procedural sedation for GI endoscopic procedures. The Obese population has a higher prevalence of obstructive sleep apnea (OSA) which is characterized by repeated obstruction of the upper airway, and leads to apnea and desaturation. This prospective, randomized study was designed to compare the effectiveness of the high flow nasal cannula and the standard nasal cannula in morbidly obese (BMI > 40) patients receiving deep intravenous sedation during colonoscopies. This study will assess whether use of the high flow nasal cannula (HFNC) leads to less intraoperative desaturation events compared to the current standard of care.

DETAILED DESCRIPTION:
The prevalence of morbid obesity is increasing worldwide. As the severity of obesity increases, the incidence of diagnosed obstructive sleep apnea also rises. Studies have shown an incidence of sleep apnea as high as 64% in patients with a body mass index (BMI) over 40 and 100% in patients with a BMI greater than 60. Patients with OSA have been shown to have significant desaturations under intravenous sedation due to airway narrowing and obstruction. Several studies have also shown that morbidly obese subjects, independent of a diagnosis of OSA, run a higher perioperative risk of adverse airway events, including hypoxia.

Many morbidly obese subjects present to our institution for GI procedures under deep sedation. Providing anesthesia for this patient population is challenging and requires careful titration of drugs and superb airway management skills. The current standard of care for oxygen delivery in this setting is a Salter nasal cannula. There are no prospective, randomized studies that compare the use of a high flow humidified nasal cannula system and standard nasal cannula in morbidly obese patients presenting for colonoscopy under anesthesia.

Humidified high flow nasal cannula (HFNC) oxygen therapy utilizes an air oxygen blend allowing from 21% to 100% FiO2 delivery and generates up to 60 L/min flow rates. The gas is heated (35 to 40 degree Celsius) and humidified through an active heated humidifier and delivered via a single limb heated inspiratory circuit (to avoid heat loss and condensation) to the subject through a large diameter nasal cannula. Theoretically, HFNC offers significant advantages in oxygenation and ventilation over conventional methods (9). Constant high flow oxygen delivery provides steady inspired oxygen fraction (FiO2) and decreases oxygen dilution. It also washes out physiologic dead space and generates positive end expiration pressure (PEEP) that augments ventilation. In the current narrative review, Sotello et al. summarized factors explained the improvement in respiratory parameters by using HFNC. (1) Washout of the nasopharyngeal dead space; (2) Reduction in inspiratory resistance associated with gas flow through the nasopharynx; (3) Improvement in respiratory mechanical parameters associated with gas temperature and state of humidification; (4) Reduction in metabolic work associated with gas conditioning; (5) Provision of mild distending pressure.

Some studies have demonstrated a positive effect of HFNC on the apnea-hypopnea index (AHI) showing that use of HFNC could decrease hypoxic episodes in subjects with repetitive upper airway obstruction such as obstructive sleep apnea. The STOP-BANG questionnaire (SB) has been used successfully to screen patients undergoing therapeutic endoscopic procedures at higher risk for sedation-related adverse events.

We are hypothesizing that the HFNC will help maintain a patent airway and improve gaseous exchange in the morbidly obese patients undergoing deep sedation for colonoscopies and will result in a significant decrease in intraoperative desaturation events, thus improving morbidity and overall safety for this subgroup.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-80
* Subjects undergoing colonoscopies
* Morbidly obese BMI ≥ 40

Exclusion Criteria:

* Subjects deemed hemodynamically unstable by the anesthesia team
* Subjects who are an aspiration risk and will require endotracheal intubation.
* Pregnancy
* Subjects with an allergy to propofol
* Patients who are unable to tolerate the high flow nasal cannula secondary to discomfort
* Subjects unwilling to sign consent
* Chronic obstructive pulmonary disease
* Patients that received medications other than lidocaine and propofol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2017-08-28 (Actual); Study Completion 2018-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Fox, MD, Study Director — University of Texas Southwestern Medical Center
Locations (2):
- United States (2):
  - Parkland Helath Hospital System, Dallas, Texas
  - Parkland Hospital, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 63 subjects consented for the study. Four subjects disqualified.
Pre-assignment Details: Four subjects disqualified due to additional procedure, induction without propofol or using fentanyl.
Period: Overall Study
Arm/Group | The High Flow Nasal Cannula | The Standard Nasal Cannula
Started | 31 | 32
Completed | 28 | 31
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | The High Flow Nasal Cannula | The Standard Nasal Cannula | Total
Number analyzed (Participants) | 28 | 31 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (7.9) | 59 (6.5) | 57 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 27 | 51
  Male | 4 | 4 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 9 | 17
  Not Hispanic or Latino | 20 | 22 | 42
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 28 | 31 | 59
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 48 (7) | 49 (10) | 49 (8.5)

OUTCOME MEASURES:

1. Primary Outcome: The Number of Desaturation Episodes
Description: The number of desaturation episodes defined as blood oxygen saturation (SpO2) below 90% during the perioperative period during colonoscopy.
Time Frame: Perioperative period during colonoscopy
Measure: Median (Inter-Quartile Range); unit: Episodes
Arm/Group | The High Flow Nasal Cannula | The Standard Nasal Cannula
Number analyzed (Participants) | 28 | 31
Episodes | 0 [0 to 1] | 0 [0 to 2]

ADVERSE EVENTS:
Time Frame: Perioperative period
Arm/Group | The High Flow Nasal Cannula | The Standard Nasal Cannula
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/31
Other Adverse Events (participants affected / at risk) | 0/28 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-22): https://cdn.clinicaltrials.gov/large-docs/62/NCT03148262/Prot_SAP_000.pdf